CLINICAL TRIAL: NCT02874170
Title: Study of the Function and Muscle Metabolism in Drepanocytose Affected Patient During a Moderate Intensity Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2014-39; 2014-A01486-41 (Other: Ansm)
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Drepanocytose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- drepanocytose affected patient (Experimental)
  Interventions: Other: Spectroscopy magnetic resonance of phosphorus 31
- Healthy volunteers (Other)
  Interventions: Other: Spectroscopy magnetic resonance of phosphorus 31

INTERVENTIONS:
Other: Spectroscopy magnetic resonance of phosphorus 31

SUMMARY:
Drepanocytose disease is the first genetic disease in the world. It results in the synthesis of an abnormal hemoglobin (HbS), which in its deoxygenated form, polymerizes and leads to structural changes of red blood cells (RBC) which then take the shape of a sickle, become more fragile, more rigid and less deformable. The fragility of GR sickle causes their mass destruction, leading to chronic anemia (i.e. low levels of GR in the blood) associated with low tissue oxygenation. More rigid and less deformable, sickle GR tend to hang in the microvessels, leading to vaso-occlusive crises (CVO) particularly painful, can cause the failure of certain organs (spleen, kidneys, brain, lung, heart, liver , bone ...) and to life-threatening patients. Preliminary studies conducted on patients with drepanocytose disease (HbSS) have demonstrated changes of muscle tissue indicating a possible failure in the supply and use of oxygen. To date, the translation of this metabolic remodeling in the muscle work is not known.

This project's main objective is to evaluate muscle function in drepanocytose attempted patients. We hypothesized that muscle remodeling associated with sickle cell disease have a functional impact on strength and muscle metabolism. The main objective is to characterize the maximal voluntary plantar flexor muscles. The criteria for these targets will be based on the comparison between healthy subjects, carriers of the sickle cell trait (HbAS) and sickle cell patients (HbSS) oxygen saturation.

The strictly non-invasive approach proposed in this project will study the functional parameters of the muscle of sickle cell disease and the possible link with the clinical manifestations of the disease, including vaso-occlusive crisis, in which tissue oxygenation and pH plays a major role.

ELIGIBILITY:
Inclusion Criteria:

* Patient affected by sickel cells and healthy volonteers presenting no contre indication to spectrometry exam.

Exclusion Criteria:

* Patient affected by hemoglobinopathies other than drepanocytose

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of phosphorus 31released during muscle exercise assesses by magnetic resonance spectroscopy | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille; Jean-Pierre MATTEI, Md, Principal Investigator — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No